CLINICAL TRIAL: NCT00245791
Title: TREATMENT OF COMPLICATED URINARY INFECTION WITH FIVE DAY HIGH DOSE LEVOFLOXACIN
Brief Title: Urinary Tract Infection Study With the Antibiotic Levofloxacin Given at a Higher Dose Over a Shorter Period of Time
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPSS-383; LOF-UTI-3
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2005-08

CONDITIONS: Complicated Urinary Infection
Keywords: Complicated Urinary Infection
MeSH Terms: interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
The purpose of the study is to compare the safety and effectiveness of the antibiotic levofloxacin by administering a higher dose of levofloxacin and using a shorter course of therapy.

DETAILED DESCRIPTION:
This study will be a pilot study of the efficacy of 750 mg of levofloxacin once daily for 5 days in the treatment of complicated urinary tract infection.

The specific objectives include:

1. To describe clinical and microbiological outcome at short and long term follow-up with 5 days levofloxacin in subjects with acute symptomatic complicated urinary infection, both with and without indwelling catheters.
2. To determine the tolerability of levofloxacin 750-mg once daily in patients with complicated urinary infection.
3. To describe some characteristics of the resolution of the inflammatory response with treatment of complicated urinary infection as demonstrated by changes in urine proteins.
4. To identify any emergence of resistant organisms in recurrent urinary infection following therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptoms of urinary infection of less than 7 days duration and an underlying structural or functional abnormality of the genitourinary tract.
2. Pre-therapy urine culture > 105 cfu/ml (> 108 cfu/L) of at least one urinary pathogen.
3. Age 18-80 years, male or female.

Exclusion Criteria:

1. Prior allergic reaction to any fluoroquinolone antimicrobial.
2. Known infection with a fluoroquinolone - resistant organism.
3. Requiring parenteral therapy because of severity of illness or unable to take oral medications.
4. Women who are pregnant or breastfeeding.
5. Requiring additional antimicrobial therapy for infections elsewhere.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-10; Study Completion 2005-07

PRIMARY OUTCOMES:
Microbiologic and clinical cure at the early post-therapy follow-up visit (12-19 days after initiating antimicrobial).

SECONDARY OUTCOMES:
Variables will include outcomes at 2 days of therapy, failure to complete therapy, adverse drug effects, long term clinical and microbiologic outcomes, and emergence of resistant organisms.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay E Nicolle, MD, FRCPC, Principal Investigator — University of Manitoba; Godfrey KP Harding, MD, FRCPC, Principal Investigator — University of Manitoba; George G Zhanel, PhD, FCCP, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - University of Manitoba, Winnipeg, Manitoba